CLINICAL TRIAL: NCT00346736
Title: Use of Acupuncture In Autistic Spectrum Disorder
Brief Title: Use of Acupuncture In Children With Autistic Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UW 04-096 T/418
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Autistic Disorder; Autism
Keywords: Alternative medicine; Traditional Chinese medicine; Acupuncture; Autistic Spectrum Disorder; Autism; Children
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture (Procedure)

SUMMARY:
Autism is a behaviorally defined, lifelong disorder of the brain, affecting at least 1-2 per 1000 children. There is an increasing trend of autism worldwide. However, to date, there is still no cure for this devastating childhood disease. Autism is characterized by deficit in language, social communication and repetitive behavior. It is estimated that the annual cost of care for autism is $13 billion in USA alone. Children with autism usually have associated behavioral problems such as aggressiveness, stereotypes, hyperactivity, emotional lability, and short attention span.

The National Institute of Child Health & Human Development and National Institute of Deafness & Communication Disorders have jointly founded the Collaborative Programs of Excellence in Autism. One of the long-term NIH goals is to develop or refine interim treatment strategy and to develop effective biological, behavioral or alternative treatment strategy for autism. There is a dire need for early identification and treatment of children with autism.

Acupuncture has been practised in China for 2 millennia. The legal status of acupuncture as a treatment technique was approved by Food & Drugs Administration in USA (1997). The therapeutic effect of acupuncture is based on stimulation at specific acupoints resulting in both local and distant effect via improving signal or modulation of electromagnetic energy. There had lack of studies of acupuncture in autism. We hope that we can study the efficacy of acupuncture in autism using clinical measurement. We hope to identify the role of acupuncture as an adjunctive treatment for autism.

DETAILED DESCRIPTION:
The aim of this study is to assess whether alternative treatment strategy such as traditional Chinese acupuncture can improve the following parameters in children with Autism (or Autistic Spectrum Disorder): cognition, communication, function and behaviour.

Randomized double-blind controlled cross-over trial in Autism: Real electro-acupuncture (R) versus Sham electroacupuncture (S)

* Subject Recruitment Parents will be informed with regard to the nature of the study, potential risks and benefits. Consent forms for enrolment, photographs/Videos taking will be obtained.
* A semi-structured diagnostic interview with the parents and neurological examination will be conducted.
* Assessment of outcomes will be performed by trained research assistant, being blinded to the treatment or control group.

Methodology:

R will consist of a total course of 12 sessions, with 3 sessions per week for 4 weeks.

* Acupuncture (AC) will be applied to specific body and scalp acupoints using sterile disposable 0.3 x 4-cm acupuncture needle (Made in China -HwaTo).
* EA instrument (Model SDZ-II Electronic Acupuncture Treatment Instrument, Suzhou China) will be connected to the handles of acupuncture needles to provide electrical stimulation for 25 minutes. No sedation is required.

S will consist of a total course of 12 sessions, with 3 sessions per week for 4 weeks.

* AC will insert into points that 5 to 10 mm away from the correct acupoint locations and maintained at a superficial level of insertion to minimize stimulation, and with the same EA.

For both R and S, electrical stimulation was monitored by an indicator light throughout the treatment period. To ensure the integrity of blinding, the acupuncturist will not discuss the acupuncture procedure with the parents or patients.

Treatment Arm (AC):

* Treatment AC for 4 weeks (3 times per week), then wash out for 2 weeks; then Sham acupuncture 3 times per week for 4 weeks

Control Arm:

* Sham acupuncture for 4 weeks (3 times per week), then wash out for 2 weeks; then Real acupuncture 3 times per week for 4 weeks

Assessment tools:

* Children will be assessed before (Week 0), washout period (Week 6) and after Treatment (Week 14).
* Control group will undergo same assessment and reassessment procedures during the same period.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled the criteria for autism of the 4th edition of the Diagnostic and Statistical Manual of Mental Disorders on the basis of observation of the child, and
* fulfilled the criteria for autism of a structured diagnostic interview of a parent using Autism Diagnostic Interview-Revised, and
* had a score on the Childhood Autism Rating Scale of 30 or more, and
* Clinical Global Impression Scale of moderately ill or markedly ill or severely ill

Exclusion Criteria:

* children on chronic anti-epileptics or neuroleptics

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-05; Primary Completion 2006-06 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavioral Checklist (ABC) will be completed by parents and teachers at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.
Ritvo-Freeman Real LIfe Scale (RFRLS) will be completed by parents and teachers at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.
Functional Independence Measure for Children (WeeFIM) will be conducted by trained Research Assistant at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.
Pediatric Evaluation Disability Inventory (PEDI) will be completed by parents and teachers at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.

SECONDARY OUTCOMES:
Leiter International Performance Scale-Revised will be conducted on patient by trained Research Assistant at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.
Reynell Language Developmental Scale will be conducted on patient by trained Research Assistant at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.
Symbolic Play Test will be conducted on patient by trained Research Assistant at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.
Clinical Global Impression Scale (CGIS) will be self administered by parent and by trained Research Assistant at Week 0, once during Week 6 to Week 7, and once during Week 14 to Week 15.

CONTACTS AND LOCATIONS:
Overall Officials: Wong Virginia, Principal Investigator — The University of Hong Kong
Locations (1):
- TWGHs Tung Wah Hospital, Hong Kong, Hong Kong